CLINICAL TRIAL: NCT00026689
Title: Evaluation for NCI Radiation Oncology Branch Clinical Research Protocols
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 000181; 00-C-0181; NCT00020280 (obsolete NCT alias)
Record Dates: First submitted 2001-11-14; First posted 2001-11-15 (Estimated); Last update posted 2019-12-12 (Actual); Status verified 2019-02-25

CONDITIONS: Prostate; Brain; Breast; Lung; Endometrial
Keywords: Evaluation; Screening; Cancer; Radiation; Eligibility
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional

GROUPS / COHORTS (1):
- 1/Cohort 1: Patients suspected of having, or with biopsy proven malignant disease or patients with a benign condition for whom radiotherapy is a potential treatment

SUMMARY:
Background:

-This protocol will provide a means for screening potential candidates for NCI Radiation Oncology Branch (ROB) protocols.

Objectives:

-To permit evaluation of patients referred to the NCI Radiation Oncology Branch in order to identify individuals who will be suitable candidates for Radiation Oncology Branch clinical research protocols.

Eligibility:

-Patients suspected of having, or with biopsy proven malignant disease or patients with a benign condition for whom radiotherapy is a potential treatment.

Design:

-This is a screening protocol. No investigational treatments will be administered on this protocol.

DETAILED DESCRIPTION:
Background:

-This protocol will provide a means for screening potential candidates for NCI Radiation Oncology Branch (ROB) protocols.

Objectives:

-To permit evaluation of patients referred to the NCI Radiation Oncology Branch in order to identify individuals who will be suitable candidates for Radiation Oncology Branch clinical research protocols.

Eligibility:

-Patients suspected of having, or with biopsy proven malignant disease or patients with a benign condition for whom radiotherapy is a potential treatment.

Design:

-This is a screening protocol. No investigational treatments will be administered on this protocol.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients suspected of having, or with biopsy proven malignant disease or patients with a benign condition for whom radiotherapy is a potential treatment.

Patient or guardian is able to provide informed consent.

EXCLUSION CRITERIA:

Candidates who do not meet the inclusion criteria.

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 903 (Actual)
Dates: Start 2000-09-11; Study Completion 2019-02-25

PRIMARY OUTCOMES:
To permit evaluation of patients referred to the NCI Radiation Oncology Branch in order to identify individuals who will be suitable candidates for Radiation Oncology Branch clinical research protocols. | Completion of study
  Evaluation of patients referred to the NCI Radiation Oncology Branch in order to identify individuals who will be suitable candidates for Radiation Oncology Branch clinical research protocols.

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States